CLINICAL TRIAL: NCT03894059
Title: Multi-Center Implementation of an Educational Program to Improve the Cardiac Arrest Diagnostic Accuracy of Ambulance Telecommunicators and Survival Outcomes for Sudden Cardiac Arrest Victims
Brief Title: An Educational Program to Improve Cardiac Arrest Diagnostic Accuracy of Ambulance Telecommunicators
Status: Active, not recruiting | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); BC Emergency Health Services (Unknown); Medacom Atlantic (Unknown); Alberta Health services (Other); Emergency Health Services Nova Scotia (Unknown); Health PEI (Unknown); Providence Health Care, British Columbia (Unknown)
Responsible Party: Sponsor
Other Study IDs: CRRF 1298
Record Dates: First submitted 2019-03-19; First posted 2019-03-28 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Heart Arrest; Heart Arrest, Out-Of-Hospital; Cardiac Arrest; Death, Sudden, Cardiac; Cardiac Arrest, Sudden; Cardiopulmonary Arrest
Keywords: cardiac arrest; bystander cardiopulmonary resuscitation CPR; dispatch-assisted CPR instructions; agonal breathing
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest; Death, Sudden, Cardiac | interventions — Early Intervention, Educational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective: Consecutive cases of out-of-hospital cardiac arrest occurring at participating sites, meeting the study eligibility criteria over a 12-month period preceding the implementation of the educational intervention for ambulance telecommunicators.
- Prospective: Consecutive cases of out-of-hospital cardiac arrest occurring at participating sites, meeting the study eligibility criteria over a 12-month period following the implementation of the educational intervention for ambulance telecommunicators.
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Other: Educational Intervention — Additional training provided to ambulance telecommunicators in participating sites to help increase recognition of agonal breathing in the presence of out-of-hospital cardiac arrest.
  Groups: Prospective

SUMMARY:
Cardiac arrest is the number one cause of death in Canada. It is often the first symptom of cardiac disease for the victims. Eighty-five percent of victims collapse in their own home. Fifty percent collapse in the presence of a family member. Bystander cardiopulmonary resuscitation (CPR) can improve the chance to survive a cardiac arrest by three to four times, but needs to be started quickly. In most communities, less than 30% of victims receive CPR before the ambulance arrives. Currently, only 8% of cardiac arrest victims can leave the hospital alive.

Many things have been tried to improve the number of times people do CPR. So far, the only thing that really increased the number of times that someone did CPR is when 9-1-1 attendants started to give CPR instructions to callers over the phone. The only problem is that about 25% of cardiac arrest victims gasp for air in the first few minutes. This can fool the 9-1-1 callers and attendants into thinking that the victim is still alive.

The investigators have looked at all the studies on how to help 9-1-1 attendants to recognize abnormal breathing over the phone. The investigators have also learned what should be taught after finishing a large survey with 9-1-1 attendants from across Canada. This survey was done with the help of psychologists and other education experts. It measured the impact of attitudes, social pressures, and 9-1-1 attendants' perceived control over their ability to recognize abnormal breathing and cardiac arrest. Then the investigators developed a teaching tool which helped Ottawa 9-1-1 attendants recognize abnormal breathing. When they could do that, they could also recognize more cardiac arrest.

The main goal of this project is to use the tool developed in Ottawa in more centres to help 9-1-1 attendants save the lives of even more cardiac arrest victims across Canada.

ELIGIBILITY:
Inclusion Criteria:

We will enroll ALL patients with prehospital cardiac arrest (absence of a detectable pulse, unresponsiveness, and apnea):

* That are of presumed cardiac origin;
* That occur in the catchment area of our participating sites; and
* For which resuscitation is attempted by a bystander and/or the emergency responders.

Exclusion Criteria:

* Cardiac arrest witnessed by paramedics after their arrival (no opportunity for bystander intervention);
* Patients younger than 16 years of age (cardiac arrest usually respiratory and rare in this population);
* Patients who are "obviously dead";
* Trauma victims, including hanging and burns; or
* Patients with cardiac arrest clearly of other non-cardiac origin including drug overdose, carbon monoxide poisoning, drowning, exsanguination, electrocution, asphyxia, hypoxia related to respiratory disease, cerebrovascular accident and documented terminal illness.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with prehospital cardiac arrest (absence of a detectable pulse, unresponsiveness, and apnea) occurring in the catchment area of any participating site during the active study period.
Sampling Method: Non-Probability Sample
Enrollment: 12224 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Change between 12 month period before and after delivery of additional education to ambulance telecommunicators
  Accessing hospital medical records or coroner's reports, assess survival of cardiac arrest victim as being discharged alive from hospital.

SECONDARY OUTCOMES:
Community Bystander Cardiopulmonary Resuscitation Rate | Change between 12 month period before and after delivery of additional education to ambulance telecommunicators
  The first member of the emergency response team to arrive at the scene will document whether or not chest compressions have been initiated by someone prior to the arrival of the emergency team.
Telecommunication-assisted CPR instructions rate | Change between 12 month period before and after delivery of additional education to ambulance telecommunicators
  By reviewing audio recordings, determine the cases where telecommunicator assistance led to delivery of chest compressions
Presence of agonal breathing | Change between 12 month period before and after delivery of additional education to ambulance telecommunicators
  Document the presence or absence of agonal breathing through review of audio recording.
Cardiac arrest recognition rate | at time of event
Time intervals | Change between 12 month period before and after delivery of additional education to ambulance telecommunicators
  call receipt to recognition of cardiac arrest, time to CPR instructions initiated

CONTACTS AND LOCATIONS:
Overall Officials: Christian Vaillancourt, MD, MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Emergency Medical Care Inc., Dartmouth, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vaillancourt C, Charette M, Naidoo S, Taljaard M, Church M, Hodges S, Leduc S, Christenson J, Cheskes S, Dainty K, Feldman M, Goldstein J, Tallon J, Helmer J, Sibley A, Spidel M, Blanchard I, Garland J, Cyr K, Brehaut J, Dorian P, Lacroix C, Zambon S, Thiruganasambandamoorthy V. Multi-centre implementation of an Educational program to improve the Cardiac Arrest diagnostic accuracy of ambulance Telecommunicators and survival outcomes for sudden cardiac arrest victims: the EduCATe study design and methodology. BMC Emerg Med. 2021 Mar 4;21(1):26. doi: 10.1186/s12873-021-00416-4. PMID 33663395